CLINICAL TRIAL: NCT00936052
Title: Phase II Pilot Trial of Hyperbaric Hyperoxygenation in Conjunction With Radiotherapy and Temozolomide In Adults With Newly Diagnosed Glioblastomas
Brief Title: Hyperbaric Hyperoxygenation With Radiotherapy and Temozolomide in Adults With Newly Diagnosed Glioblastoma
Acronym: HBO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurological Surgery, P.C. (Other)
Responsible Party: J. Paul Duic, MD, Long Island Brain Tumor Center at Neurological Surgery, P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIBTC-2008-2
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Glioblastomas; Gliosarcoma
Keywords: glioblastomas; GBM; gliosarcoma; blastoma; sarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Sarcoma | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — in addition to standard radiation and chemotherapy, you will also receive the experimental hyperbaric treatment prior to each radiation treatment (Monday-Friday) during the initial six weeks of treatment. Prior to the first hyperbaric treatment. The hyperbaric treatment lasts approximately thirty minutes. During the hyperbaric treatment, the participant will lie on a stretcher in the hyperbaric chamber and breathe oxygen at greater than normal atmospheric pressure. The investigator will monitor the increased oxygen levels in the tissue by placing a noninvasive electrode on your skin. After each hyperbaric treatment, we will measure your blood sugar by finger-stick to check for hypoglycemia (low blood sugar). If detected, hypoglycemia will be treated by standard medical measures.
  Other Names: Oxygenation; oxygen tank

SUMMARY:
Standard treatment for glioblastomas includes radiation and chemotherapy with a drug called temozolomide (Temodar); however, glioblastomas frequently develop resistance to standard treatment and recur or progress. Glioblastomas are known to have decreased levels of oxygen compared to normal tissues. There is evidence that these lower oxygen levels in glioblastomas may contribute to their ability to resist treatment effects of radiation and chemotherapy. In this study we will look to increase the oxygen concentration within the glioblastoma by adding hyperbaric treatments (the experimental part of this study) to standard treatment with radiation and temozolomide in order to see whether increasing the oxygen concentration within the tumor increases the tumor-killing ability of standard radiation and chemotherapy.

In addition, the investigators are interested to evaluate the effect of this treatment protocol on a person's quality of life and level of stress, and, therefore, the investigators will ask subjects to complete several brief questionnaires while they are on-study.

DETAILED DESCRIPTION:
All enrolled study subjects will receive treatment. Nobody will receive placebo. Before starting on-study, the investigators require standard blood tests (blood counts, chemistries, liver function tests, etc), urinalysis, serum pregnancy test (females of childbearing potential only) and an MRI with contrast (or CAT scan if you are unable to obtain MRI) that the investigators routinely obtain before starting any new treatment or chemotherapy.

Standard treatment for newly diagnosed glioblastomas after surgery begins with six weeks of combined radiation (Monday-Friday) and chemotherapy with an oral drug called temozolomide (Temodar) that patients normally take at home daily (including weekends) during the six weeks. Patients then have four weeks off treatment. After four weeks off, patients resume taking temozolomide on a monthly basis. During this phase of treatment, patients take a higher dose of temozolomide for only five days out of every twenty eight days (they take the drug only during the first five days of every 28 day cycle with the remaining 23 days off drug). Patients continue taking temozolomide on a monthly basis until tumor progression, they complete six to twelve months of treatment or they are unable to tolerate the drug any longer due to side effects.

Temozolomide is typically taken once daily on an empty stomach one-half hour after taking an anti-nausea medication that is also prescribed by your physician. Patients taking temozolomide are also instructed to take lactulose as needed for constipation.

During the initial six weeks of combined radiation and chemotherapy, patients also take an antibiotic to protect against a specific type of pneumonia that commonly occurs in people with weakened immune systems (pneumocystis carinii). Following completion of the combined phase of radiation and chemotherapy, continuation of the antibiotic depends upon the discretion of the treating physician.

In this study, in addition to standard radiation and chemotherapy described above, the patient will also receive the experimental hyperbaric treatment prior to each radiation treatment (Monday-Friday) during the initial six weeks of treatment. Prior to the first hyperbaric treatment, the patient will need to have a chest x-ray performed to make certain that you do not have any preexisting abnormal air spaces in the chest or lungs that could be worsened by hyperbaric treatment. The hyperbaric treatment lasts approximately thirty minutes. During the hyperbaric treatment, the patient will lie on a stretcher in the hyperbaric chamber and breathe oxygen at greater than normal atmospheric pressure. The investigators will monitor the increased oxygen levels in the tissue by placing a noninvasive electrode on your skin. After each hyperbaric treatment, the investigators will measure the participants blood sugar by finger-stick to check for hypoglycemia (low blood sugar). If detected, hypoglycemia will be treated by standard medical measures.

Blood tests will be obtained as per routine standard of care (weekly during the initial six weeks of combined radiation and chemotherapy) and on days # 21 and 28 (+/- 2 days) of each cycle of monthly temozolomide.After the initial MRI (or CAT scan), subsequent MRI's (or CAT scans) will be obtained per standard of care: four weeks after completion of radiation and then generally after every two cycles of chemotherapy unless medically indicated at other time points.

Other scans such as PET scans may be obtained if medically indicated as per standard of care.

This study also looks to evaluate the effect of this treatment regimen on the quality of life for the patient and level of stress. Therefore, the investigators will ask the patient to complete three brief questionnaires at several different time points: before starting the study, at the follow-up visit three to four weeks after completion of radiation, after completion of every two cycles of monthly temozolomide and after coming off study (if possible.) The patient will remain on study until completion of one year of treatment, the patient may voluntarily elect to withdraw from study, the patient cannot tolerate further treatment or side effects prevent continuing on study or there is evidence of tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than/equal to 18 years old;
2. histologically confirmed newly diagnosed WHO IV glioblastoma/gliosarcoma;
3. Subjects are eligible postoperatively following biopsy, subtotal or gross total resection with or without radiographic evidence of residual disease;
4. recent contrast-enhanced MRI within 4 weeks of enrollment onto protocol;
5. no prior or concurrent antitumor therapy;
6. Karnofsky performance score >= 60;
7. no significant comorbidities;
8. signed informed consent;
9. adequate bone marrow function;
10. adequate liver and renal function;
11. males, females and minorities are eligible without any preference to gender or race;
12. negative serum pregnancy test.

Exclusion Criteria:

1. Greater than/equal to 18 years old;
2. histologically confirmed newly diagnosed WHO IV glioblastoma/gliosarcoma;
3. Subjects are eligible postoperatively following biopsy, subtotal or gross total resection with or without radiographic evidence of residual disease;
4. recent contrast-enhanced MRI within 4 weeks of enrollment onto protocol;
5. no prior or concurrent antitumor therapy;
6. Karnofsky performance score >= 60;
7. no significant comorbidities;
8. signed informed consent;
9. adequate bone marrow function;
10. adequate liver and renal function;
11. males, females and minorities are eligible without any preference to gender or race;
12. negative serum pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
to generate preliminary data of the anti-tumor efficacy of hyperbaric oxygenation in conjunction with radiotherapy and chemotherapy,to determine median progression-free survival, to determine median survival and to determine median 2 year survival. | one year

SECONDARY OUTCOMES:
to determine the health related quality of life of this treatment regimen and its influence upon subjects'' perceived level of traumatic stress throughout the course of treatment. | one year

CONTACTS AND LOCATIONS:
Overall Officials: J Paul Duic, MD, Principal Investigator — Long Island Brain Tumor center at Neurological Surgery P.C.; Jai Grewal, MD, Principal Investigator — Long Island Brain Tumor Center at Neurological Surgery P.C.
Locations (2):
- United States (2):
  - Long Island Brain Tumor Center at Neurological surgery P.C., Commack, New York
  - Long Island Brain Tumor Center at Neurological Surgery P.C., Great Neck, New York